CLINICAL TRIAL: NCT05577182
Title: A Phase 1, Open-Label, Multicenter Study of INCA32459 in Participants With Select Advanced Malignancies
Brief Title: Study of INCA32459 a LAG-3 and PD-1 Bispecific Antibody in Participants With Select Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCA 32459-101; 2022-501505-13-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignancies
Keywords: LAG-3; bispecific antibody; melanoma; squamous cell carcinoma of the head and neck (SCCHN)
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Part 1 will be dose escalation using a statistical hybrid design to identify the RDE(s). Part 2 will be dose expansion portion which will administer the RDE(s) defined in Part 1 to participants in 2 tumor-specific cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation (Experimental): INCA32459 will be administered at a protocol defined starting regimen intravenously. Subsequent dose regimens will be determined during study conduct.
  Interventions: Drug: INCA32459-101
- Part 2: Dose Expansion Cohort Disease Group 1 (Experimental): INCA32459 will be administered at the recommended dose or doses for expansion (RDE[s]) for unresectable or metastatic melanoma.
  Interventions: Drug: INCA32459-101
- Part 2: Dose Expansion Cohort Disease Group 2 (Experimental): INCA32459 will be administered at the recommended dose or doses for expansion (RDE[s]) for recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) that is PD-L1 positive.
  Interventions: Drug: INCA32459-101

INTERVENTIONS:
Drug: INCA32459-101 — solution for infusion

SUMMARY:
This is a multicenter, open-label, single-arm study to investigate the safety, tolerability, PK, pharmacodynamics and preliminary activity of INCA32459 in participants with selected advanced malignancies. Part 1 (dose escalation) will determine the recommended dose of INCA 32459 for expansion (RDE) and the maximum tolerated dose (MTD). Part 2 (dose expansion) will further evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary antitumor activity of INCA 32459 at the recommended dose(s) for expansion in 2 tumor-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced malignancies as follows:

  1. Part 1 only: Participants with the select advanced malignancies as specified in the protocol.
  2. Part 2 only:

     * Cohort 1 only: Participants with Stage III (unresectable) or Stage IV (metastatic) melanoma that is considered nonamenable to curative treatments or procedures.
     * Cohort 2 only: Participants with histologically or cytologically confirmed recurrent/metastatic SCCHN that is PD-L1 positive (CPS ≥ 1) which is not amenable to local therapy with curative intent.
* Participants must have experienced disease progression after treatment with standard therapies, or are intolerant to or ineligible for standard treatment:

  1. Part 1: All available standard therapies, including anti-PD-(L)1 and platinum-based therapy, if applicable, that are known to confer clinical benefit. Prior anti-PD-(L)1 therapy should not have been discontinued because of intolerance.
  2. Part 2: Available standard therapies, including anti-PD-(L)1 and platinum-based therapy, if applicable, that are known to confer clinical benefit. Prior anti-PD-(L)1 therapy should not have been discontinued because of intolerance. Part 2 participants may have received up to 2 prior systemic therapies in the a advanced/metastatic setting.
* ECOG performance status of 0 or 1
* Part 2 only: Measurable disease according to RECIST v1.1.
* Part 2 only: Willingness to undergo a fresh tumor biopsy at screening (core or excisional).
* Part 2 only: Willingness to undergo a fresh tumor biopsy at screening and on-treatment in selected participant.
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Prior treatment with any LAG-3- or MHC Class II-directed therapy for current malignancy, or any prior malignancy.
* Treatment with anticancer therapies or participation in another interventional clinical study within 28 days before the first administration of study treatment (this includes curative radiation to the thorax or systemic anticancer therapies).
* Not recovered to ≤ Grade 1 or baseline from residual toxicities of prior therapy (with exceptions specified in the protocol).
* Not recovered adequately from toxicities and/or complications from surgical intervention before starting study treatment.
* Palliative radiation therapy administered within 1 week of first dose of study treatment or radiation therapy in the thoracic region that is > 30 Gy within 6 months of the first dose of study treatment.
* Any known additional malignancy that is progressing or requires active treatment; history of other malignancy within 3 years of the first dose of study treatment (with exceptions specified in the protocol).
* Evidence of interstitial lung disease or history of interstitial lung disease, or active, noninfectious pneumonitis.
* Active autoimmune disease requiring systemic immunosuppression with corticosteroids (> 10 mg/day of prednisone or equivalent) or immunosuppressive drugs within 2 years before the first dose of study treatment.
* Untreated brain or CNS metastases or brain or CNS metastases that have progressed (eg, evidence of new or enlarging brain metastasis or new neurological symptoms attributable to brain or CNS metastases).
* Chronic treatment with systemic steroids (> 10 mg/day of prednisone or equivalent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Part 1: Occurrence of Dose Limiting Toxicities (DLTs) | Up to approximately 12 months
  Toxicities occurring during Part 1 will define tolerability. DLTs will be assessed for severity by the investigator using CTCAE v5.0 criteria.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to approximately 12 months
  TEAE is any Adverse Event (AE) either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Number of Participants with Dose Interruptions due to TEAE | Up to approximately 12 months
  Dose interruptions will occur according to protocol guidelines.
Number of Participants discontinue study due to TEAE | Up to approximately 12 months
  TEAE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 12 months
  Defined as having Complete Response (CR) or Partial Response (PR), as determined by the investigator by radiographic disease assessment according to RECIST v1.1 or Lugano criteria (B-cell lymphomas only).
Disease Control Response (DCR) | Up to 12 months
  Defined as having CR, PR, or Stable Disease (SD) as determined by the investigator by radiographic disease assessment according to RECIST v1.1. or Lugano criteria (B-cell lymphomas only).
Duration of Response (DOR) | Up to 12 months
  Defined as the time from earliest date of disease response (Completed Response or Partial Response) until earliest date of disease progression as determined by the investigator by radiographic disease assessment according to RECIST v1.1 or Lugano criteria (B-cell lymphomas only) or death due to any cause if occurring sooner than progression.
PK parameters: Cmax | Up to 24 months
  Defined as the maximum (peak) plasma drug concentration
PK parameters: tmax | Up to 24 months
  Defined as the time to reach maximum (peak) plasma concentration following drug administration
PK parameters: Cmin | Up to 24 months
  Defined as concentration at the end of the dosing interval
PK Parameters: AUC | Up to 24 months
  Defined as the area under the plasma concentration-time curve
PK Parameters: CL | Up to 24 months
  Defined as the apparent total body clearance of the drug from plasma
PK Parameters: Vz | Up to 24 months
  Defined as apparent volume of distribution during terminal phase
PK Parameters: t1/2 | Up to 24 months
  Defined as Elimination half-life (to be used in one-or noncompartmental model)
Receptor Occupancy | Up to 24 months
  Defined as PD-1 receptor occupancy in peripheral blood samples.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (2):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Texas Md Anderson Cancer Center, Houston, Texas
- Belgium (5):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Chu Ucl Namur University Hospital Mont-Godinne, Yvoir
- Centro Ricerche Cliniche Di Verona (Crc), Verona, Italy
- Spain (5):
  - Hospital Quironsalud Barcelona, Barcelona
  - Ico Institut Catala D Oncologia, L'Hospitalet de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: No